CLINICAL TRIAL: NCT07153965
Title: An Open-label, Single-arm, Multicenter Phase II Study of Sacituzumab Tirumotecan (Sac-TMT) Plus Tagitanlimab in Previously Treated PD-L1-positive Locally Advanced or Metastatic Triple Negative Breast Cancer (TNBC)
Brief Title: Sacituzumab Tirumotecan Plus Tagitanlimab in Previously Treated Locally Advanced or Metastatic Triple Negative Breast Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SKB264-IIT-017
Record Dates: First submitted 2025-08-24; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Triple Negative Breast Cancer (TNBC); PD-L1 Positive
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- sac-TMT plus Tagitanlimab (Experimental)
  Interventions: Drug: Sacituzumab Tirumotecan plus Tagitanlimab

INTERVENTIONS:
Drug: Sacituzumab Tirumotecan plus Tagitanlimab — Sacituzumab Tirumotecan 5mg/kg intravenously (IV) infusion every 2 weeks on Day 1, Tagitanlimab 900mg IV every 2 weeks on Day 1, until disease progression, unacceptable toxic effects, withdrawal from the trial, or death, whichever occurred first.

SUMMARY:
This is an open-label, single-arm, multicenter phase II study to evaluate the safety and efficacy of sac-TMT plus Tagitanlimab in patients with PD-L1-positive locally advanced or metastatic TNBC.

ELIGIBILITY:
Key inclusion criteria include but are not limited to:

* Age ≥ 18 years at the time of signing informed consent.
* Histologically and/or cytologically confirmed triple-negative breast cancer (TNBC) based on the most recent biopsy or other pathological specimens, including:

  1. Definition of human epidermal growth factor receptor 2 (HER2) negative: immunohistochemistry (IHC) of 0 or 1+; if HER2 is 2+ by IHC, negative HER2 expression must be confirmed by fluorescencein situ hybridization (FISH); Estrogen and progesterone receptor negative means that less than 1% of the cells express hormone receptors as indicated by IHC.
  2. Tumor stage: locally advanced, recurrent, or metastatic TNBC; locally advanced cases must be confirmed by the investigator as unsuitable for curative surgical resection.
* Patients with unresectable locally advanced or metastatic triple-negative breast cancer:

  1. Those who have received chemotherapy combined with a PD-(L)1 inhibitor as first-line treatment for locally advanced or metastatic disease and experienced progression ≥ 3 months later.
  2. Those who received chemotherapy combined with a PD-(L)1 inhibitor in the neoadjuvant and/or adjuvant setting and experienced recurrence or disease progression to unresectable locally advanced or metastatic disease ≥ 3 months later but within 12 months.
  3. Those who received chemotherapy combined with a PD-(L)1 inhibitor in the neoadjuvant and/or adjuvant setting and experienced recurrence or disease progression to unresectable locally advanced or metastatic disease after ≥ 12 months, and have subsequently progressed on first-line treatment for locally advanced or metastatic disease.
* Newly diagnosed brain metastases at screening must be stable for ≥ 4weeks after local treatment (e.g., radiotherapy) with imaging confirmation.
* The most recent tumor tissue sample from the primary and/or metastatic lesion must show a PD-L1 combined positive score (CPS) ≥ 1.
* Patients must have at least one measurable lesion per RECIST v1.1 criteria; those with only skin or bone lesions cannot be included.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to1.
* Patients must have adequate organ and bone marrow function (no blood transfusion, recombinant human thrombopoietin, or colony stimulating factor therapy has been received within 2 weeks prior to the treatment)
* Patients of childbearing potential (male or female) must use effective medical contraception from consent until 6 months after the end of the dosing period.

Key exclusion criteria include but are not limited to:

* Previously received any of the following treatments (including in the adjuvant or neoadjuvant setting):

  1. Targeted TROP2 therapy.
  2. Any drug treatment targeting topoisomerase I, including antibody drug conjugates (ADC) therapy.
* Known to have meningeal metastasis, brainstem metastasis, spinalcord metastasis, and/or compression, active central nervous system(CNS) metastasis. Patients with previously treated brain metastases canparticipate if clinically stable for at least 4 weeks before dosing and do not require corticosteroids or anticonvulsants for at least 14 days. Patients with untreated asymptomatic brain metastases must require investigator approval.
* Has a history of documented severe dry eye syndrome, severe Meibomian gland disease and/or blepharitis, or corneal disease that prevents/delays corneal healing.
* Within 3 years before administration having other malignancies (except forthose cured by local treatment, such as basal cell carcinoma of the skin,squamous cell carcinoma of the skin, cervical carcinoma in situ, etc.).
* Has uncontrolled, significant cardiovascular disease or risk factors, uncontrollable systemic diseases.
* Presence of steroid-requiring (non-infectious) interstitial lung disease (ILD)or a history of non-infectious pneumonia, currently having ILD or non-infectious pneumonia, or suspected ILD or non-infectious pneumonia that cannot be ruled out by imaging at screening.
* Unresolved toxicities from previous anti-tumor therapy to ≤ Grade 1 (based on NCI CTCAE v5.0) or the level specified in the inclusion and exclusion criteria.
* Patients with active chronic inflammatory bowel disease, gastrointestinal obstruction, severe ulcers, gastrointestinal perforation, abdominal abscess, or acute gastrointestinal bleeding.
* Having an active autoimmune disease requiring systemic treatment inthe past two years.
* Known active tuberculosis, hepatitis B or hepatitis C.
* Human Immunodeficiency Virus (HIV) test positive or history of Acquired Immunodeficiency Syndrome (AIDS); known active syphilis infection.
* Known allergy to the study drug or any of its components, known history of severe hypersensitivity to other biological products
* Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) as Assessed by Investigator per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) | up to approximately 60 months
  ORR is defined as the proportion of participants who achieve a complete response (CR) or partial response (PR) that is confirmed at least 4 weeks after initial documentation of response.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) as Assessed by Investigator per RECIST Version 1.1 | up to approximately 60 months
  PFS is defined as time from date of randomization until the date of first objective progressive disease (PD) by investigator assessment according to RECIST v1.1 or death from any cause, whichever comes first.
Overall Survival (OS) | up to approximately 60 months
  OS is defined as the time from randomization until the date of death from any cause.
Disease control response (DCR) as Assessed by Investigator per RECIST Version 1.1 | up to approximately 60 months
  DCR is defined as the proportion of participants who achieve a complete response (CR), partial response (PR) or or stable disease (SD) .
Duration of response (DoR) | up to approximately 60 months
  DoR is defined as the time from the first objective response (CR/PR) to the first documented disease progression (PD) according to RECIST v1.1 or death from any cause, whichever comes first.
Safety and Tolerability | up to approximately 60 months
  Incidence and severity of AEs and SAEs (per CTCAE 5.0)
Health-related quality of life (HRQoL) evaluated using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) | up to approximately 60 months
  Mean change from baseline in the EORTC QLQ-C30
Health-related quality of life (HRQoL) evaluated using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Breast Cancer Module 23 (EORTC QLQ-BR23) | up to approximately 60 months
  Mean change from baseline in the EORTC QLQ-BR23

OTHER OUTCOMES:
TROP2, PD-L1, tumor-infiltrating lymphocytes (TILs), lymphocyte subpopulation | up to approximately 60 months
  Explore potential biomarkers that predict the treatment response and prognosis of TNBC, including but not limited to the expression levels of TROP2, PD-L1, tumor-infiltrating lymphocytes (TILs), lymphocyte subpopulation.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China